CLINICAL TRIAL: NCT05600751
Title: Radiosurgery of Ganglion StELlatum In Patients With REFractory Angina Pectoris
Acronym: RELIEF-AP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Collaborators: Nemocnice AGEL Trinec-Podlesi a.s. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RELIEF-AP Trial
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Myocardial Ischemia
Keywords: radiosurgery; ganglion stellatum; angina pectoris; coronary artery disease; myocardial ischemia
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiosurgery of Ganglion Stellatum (Experimental): Patients will undergo radiosurgery of the ganglion stellatum (left one or both)
  Interventions: Procedure: Radiosurgery of ganglion stellatum

INTERVENTIONS:
Procedure: Radiosurgery of ganglion stellatum — Patients will undergo radiosurgery of ganglion stellatum (left one or both)

SUMMARY:
The core hypothesis to be tested is that the radiosurgery of stellate ganglion (left one or both if left-sided without full relief of symptoms) is an effective therapy of refractory angina pectoris in patients with no other therapeutic options - proof of concept study.

DETAILED DESCRIPTION:
Design: prospective, interventional trial (University Hospital Ostrava, Cardiocentre AGEL Podlesi Hospital Trinec)

* radiosurgery of left GS after confirmation of responding to anesthetic blockade
* in case of remaining AP after three months, radiosurgery of right GS in case of response confirmation to anesthetic blockade (patients must be responders of anesthetic blockade of left stellate ganglion)
* Seattle Angina Questionary (SAQ) and amount of nitrate usage for responding confirmation
* Radiotherapy 40 Gy
* 2-year follow-up
* Scheduled follow-up visits: 1, 3, 6, 12, and 24 months (24)

Preliminary examination: selective coronary angiography, transthoracic echocardiography, stress test, 6 min walk test, SAQ (19-item)

Endopoints:

Primary Endpoints: SAQ, safety of the radiosurgery of GS Secondary Endpoints:usage decrease of angina relief drugs, 6 min walk test improvement

Follow-up visits examination, Restage: 6 min walk test, SAQ, amount of nitrate usage, ECG, blood tests incl. NT-proBNP, NSE

ELIGIBILITY:
Inclusion Criteria:

* Patients must have coronary artery disease (CAD) with refractory angina pectoris (AP).
* Patients must have a maximum of tolerated medication therapy of angina pectoris available.
* Patients must have done the maximum possible revascularization of CAD.
* Two certificated independent interventional cardiologists and two cardiac surgeons must conclude that further revascularization (including CABG) is not possible/not effective/ with high risk.
* Age ≥ 18 years.
* Patients must have any stress test with proof of myocardial ischemia (dobutamine echocardiography, gated Tc-SPECT of myocardium).
* Life expectancy at least 24 months (not limited due to severe comorbidities)
* Patients must be responders of anesthetic blockade of the left stellate ganglion (GS) - clinically significant relief of AP symptoms after blockade at least twice.
* Patients must provide verbal and written informed consent to participate in the study.

Exclusion Criteria:

* Life expectancy less than 24 months
* Non-responders of anesthetic blockade of GS
* Impossibility to undergo a stress test.
* Myocardial infarction in last 4 weeks
* Heart failure - class IV NYHA
* Unwillingness to participate or inability to comply with the protocol for the duration of the study
* Patients who are pregnant, and patients with reproductive capability will need to use adequate contraception during the time of participation in the study
* History of radiotherapy in the head and neck region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Seattle Angina Questionnaire | 24 months
  The Seattle Angina Questionnaire is a cardiac disease-related quality-of-life measure with 19 items. A lower score corresponds to a lower level of functioning. The scores are classified as "minimal (scores 75-100), mild (50-74), moderate (25-49), and severe (0-24).
Safety of radiosurgery of ganglion stellatum | 24 months
  Safety of radiosurgery of ganglion stellatum will be observed and assessed according to the occurrence of adverse events

SECONDARY OUTCOMES:
Usage of angina pectoris relief drugs | 24 months
  The change of angina pectoris relief drugs will be evaluated
Six-minute walk test improvement | 24 months
  Change in the six-minute walk test will be evaluated before and after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Cvek, Assoc.Prof.,MD,Ing.,PhD, Principal Investigator — University Hospital Ostrava
Locations (2):
- Czechia (2):
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - AGEL Podlesí Hospital Třinec, Třinec, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: No
Individual participant data may be made available upon request.